CLINICAL TRIAL: NCT05839106
Title: A Phase I/IIa Study to Evaluate the Tolerance, Safety, Pharmacokinetic Characteristics and Preliminary Efficacy of PM1032 in Patients With Advanced Solid Tumors
Brief Title: Phase I/IIa Study for PM1032 in the Treatment of Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PM1032-AB001M-ST-R
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Advanced Tumor
Keywords: CLDN 18.2; 4-1BB

STUDY DESIGN:
Intervention Model Description: In dose escalation stage, three subjects will be enrolled at the protocol starting dose of PM1032 for 21 Days DLT observation, followed by same dose every 2 weeks (Q2W) until they meet the discontinuation criteria.
  Dose escalation will proceed to the next dose level according to the 3+3 design.
  Dose expansion stage of the study will be initiated at the Sponsor's discretion at the dose level and treatment schedule which was established as the recommended Phase 2 dose (RP2D) in the dose escalation stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM1032 monotherapy (Experimental): PM1032 0.3mg/kg-12mg/kg
  Interventions: Drug: PM1032 injection

INTERVENTIONS:
Drug: PM1032 injection — Subjects will receive PM1032 by intravenous administration.
  Other Names: PM1032

SUMMARY:
The study is being conducted to evaluate safety, tolerability, pharmacokinetics and preliminary efficacy of PM1032 for patients with advanced tumors, also to explore the recommended Phase Ⅱ Dose（RP2D） of PM1032.

DETAILED DESCRIPTION:
PM1032 is a Bispecific Antibody Targeting CLDN18.2 and 4-1BB.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in clinical study; fully understand the study and sign informed consent voluntarily;
* Male or female aged 18 to 75 years;
* Subjects with malignant tumor confirmed by histology or cytology, subjects with advanced malignant solid tumors who have no standard treatment, have failed standard treatment or are not eligible for standard treatment:

  1. Phase I dose escalation stage: gastric/gastroesophageal junction adenocarcinoma, esophageal cancer, etc.;
  2. Phase I dose expansion stage, phase IIa dose expansion stage: gastric/gastroesophageal junction adenocarcinoma, esophageal cancer, other tumors; CLDN18.2-positive tumor expression as determined by the CLDN18.2 IHC assay in central laboratory.
* Adequate organ function;
* ECOG score was 0-1;
* Expected survival≥12 weeks;

Exclusion Criteria:

* History of severe allergic, severe allergy to drugs or known allergy to any component of the drug in this study;
* Previous exposure to immune co-stimulatory molecule agonists such as 4-1BB mono/bispecific antibodies, etc;
* Patients who received CLDN18.2-targeted mono/bispecific antibodies or cell therapy;
* Cerebral parenchymal metastasis or meningeal metastasis with clinical symptoms were deemed unsuitable for this study by the investigator;
* Current definite interstitial lung disease or non-infectious pneumonitis, except for local radiotherapy;
* Current presence of uncontrolled pleural, pericardial, and peritoneal effusions;
* Adverse reactions to previous anti-tumor therapy have not recovered to NCI-CTCAE V5.0 rating≤1;
* Patients ever received the following treatments or drugs prior to the study treatment:

  1. Major organ surgery within 28 days prior to initiation of trial treatment or requiring elective surgery during the trial period;
  2. Received live attenuated vaccine within 28 days prior to the study treatment;
  3. Received chemotherapy, radical/extensive radiation, biotherapy, endocrine therapy and other anti-tumor drug therapy within 4 weeks of the first administration;
  4. Received systemic glucocorticoid or other immunosuppressive therapy within 2 weeks before the trial treatment;
* Active bleeding within 3 months of the first administration;
* History of allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation;
* Pregnant or lactating women;
* Other conditions considered unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity（DLT） | up to 21 days
  Occurrence of DLT after receiving PM1032 injection
Assess the incidence and severity of treatment-related adverse events | Up to 30 days after last treatment
  The incidence and severity of treatment-emergent adverse events (TEAEs) and treatment related adverse events (TRAEs) graded according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Principal Investigator — Shanghai Orient Hospital
Locations (3):
- China (3):
  - Shulan (Hang Zhou) Hospital, Hangzhou
  - The first affiliated hospital of nanchang university, Nanchang
  - Shanghai Orient Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract, articles or papers) or maked any presentations.
Time Frame: after the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.